CLINICAL TRIAL: NCT05063097
Title: Assessment of ADDICTion to Psychoactive Drug Use in Intensive Cardiac Care Units - The ADDICT-CCU Study
Brief Title: Addiction in Intensive Cardiac Care Units
Acronym: ADDICT-CCU
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Coeur et Recherche (Unknown)
Responsible Party: Sponsor
Other Study IDs: APHP190870; 2021-A00702-39 (Other: ANSM - IDRCB)
Record Dates: First submitted 2021-07-19; First posted 2021-09-30 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Intensive Care Unit Syndrome; Drug Abuse; Substance-Related Disorders; Cardiovascular Events; Cardiac Disease
Keywords: Prevalence; Drug Abuse; Illicit drug use; Substance-Related Disorders; Intensive cardiac care unit; Cannabis; Cocaine; Cardiovascular events; Psychoactive drug use
MeSH Terms: conditions — Substance-Related Disorders; Heart Diseases; Marijuana Abuse | interventions — Urinalysis; Weights and Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CCU patients: All consecutive patients over 18 years admitted to the CCU.
  Interventions: Other: urine test; Other: Fagerström questionnaire; Other: Exhaled carbon monoxide (CO) measurement

INTERVENTIONS:
Other: urine test — The following illicit drugs will be evaluated for all consecutive patients by urine drug assay (NarcoCheck®, Kappa City Biotech SAS, Montluçon, France) within two hours of admission to the ICCU: i) cannabinoids (tetrahydrocannabinol [THC]), including cannabis and hashish; ii) cocaine and metabolites, including cocaine and crack; iii) amphetamines; iv) MDMA; and v) heroin and other opioids. In addition to the analysis of psychoactive drug use, the investigators will also use the NarcoCheck® urine drug assay to evaluate the associated use of the following psychostimulant drugs: barbiturates, benzodiazepines, tricyclic antidepressant drugs, methadone and buprenorphine.
Other: Fagerström questionnaire — Tobacco consumption will also be evaluated for each patient using a Fagerström questionnaire.
Other: Exhaled carbon monoxide (CO) measurement — Active smoking will also be systematically investigated in all patients using a standardized exhaled carbon monoxide (CO) measurement with a CO-Check Pro device (Bedfont Scientific Ltd, Kent, UK) on arrival, with a measure of > 3 parts per million (ppm) signifying active smoking.

SUMMARY:
Background:

Illicit drug use is a growing issue in Europe and leading cause of acute cardiac events in patients admitted to intensive cardiac care units. Indeed, cardiovascular complications are one of the main causes of death due to illicit drug use. However, its prevalence in patients hospitalized in intensive cardiac care units is unknown.

Objectives:

This large multicenter prospective study will assess the prevalence of illicit drug use in consecutive patients hospitalized in intensive cardiac care units by urine drug assay.

Eligibility:

* Patient over 18 years old admitted to intensive Cardiac Care Unit (CCU) for any reason.
* Without hospitalization for a planned interventional procedure.
* Without hospitalization for more than 24 hours at any hospital facility before admission to the CCU.

Design:

* Multicentre cohort study with a prospective enrolment of all consecutive patients admitted to the CCU to assess the prevalence of illicit drug use in 40 centers throughout France.
* Participants will be screened with a physical exam, medical history and addiction survey.
* Participants will be screened for drug use by urine drug assay (NarcoCheck®, Kappa City Biotech SAS, Montluçon, France) and for tobacco by standardized exhaled carbon monoxide (CO) measurement with a CO-Check Pro device (Bedfont Scientific Ltd, Kent, UK).
* Participants will be followed at 6 months of follow-up to assess the occurrence of cardiovascular events.

DETAILED DESCRIPTION:
Objective:

Illicit drug use is a growing issue in Europe. In France, the prevalence of the illicit use of any drug is 11.4% of the population, ahead of Italy (10.6%), the United Kingdom (8.7%) and Germany (7.8%).

Cardiovascular complications are one of the main causes of death due to psychoactive drug use with more than 100,000 deaths per year are due to psychoactive drug use in France. Although the use of illicit drugs may be involved in several acute cardiac events in patients admitted to intensive cardiac care units (CCU), its prevalence in patients hospitalized in CCU is unknown. Interestingly, the current guidelines recommend only a declarative survey to investigate psychoactive drug use but no systematic urine or plasma screening. However, the rate of underreporting of these illegal substances remains high. To our knowledge, no study has ever consecutively assessed the prevalence of psychoactive drug use using systematic urine or plasma screening at the time of CCU admission. Because illicit drug use is a potential cardiovascular risk factor, accurate drug screening may initiate addictology management, modify the treatment and improve patient prognosis after a cardiovascular event.

The aim of the prospective ADDICT-CCU study is to assess the prevalence of illicit drug use in consecutive patients hospitalized in intensive cardiac care units by urine drug assay.

Study population:

All consecutive patients over 18 years admitted to the CCU during a 3 week recruitment period in 40 centers. The main exclusion criteria will be hospitalization for a planned interventional procedure, dementia, or hospitalization for more than 24 hours at any hospital facility before admission to the CCU. Informed consent will be obtained from all participants.

Design:

The investigators will conduct a multicentre cohort study with a prospective enrolment of all consecutive patients admitted to the CCU to assess the prevalence of psychoactive drug use in 40 centers throughout France. Anonymized data supporting the findings of this study will be collected using CleanwebTM software.

Outcome Measures:

The primary outcome will be the prevalence of at least one illicit drug among all consecutive patients hospitalized in the CCU.

The following psychoactive drugs will be evaluated for all consecutive patients by urine drug assay (NarcoCheck®, Kappa City Biotech SAS, Montluçon, France) within two hours of admission to the CCU: i) cannabinoids (tetrahydrocannabinol [THC]), including cannabis and hashish; ii) cocaine and metabolites, including cocaine and crack; iii) amphetamines; iv) MDMA; and v) heroin and other opioids.

In addition to the analysis of illicit drug use, the investigators will also use the NarcoCheck® urine drug assay to evaluate the associated use of the following psychoactive drugs: barbiturates, benzodiazepines, tricyclic antidepressant drugs, methadone and buprenorphine. Tobacco consumption will also be evaluated for each patient using a questionnaire with three choices: "never smoked," "smoking cessation" specifying the number of years, or "active smoking." Active smoking will also be systematically investigated in all patients using a standardized exhaled carbon monoxide (CO) measurement with a CO-Check Pro device (Bedfont Scientific Ltd, Kent, UK) on arrival, with a measure of > 3 parts per million (ppm) signifying active smoking. Every patient will be provided with relevant instructions regarding the urine drug assay and exhaled CO measurement, and trained investigators will conduct the tests.

Regarding the secondary outcomes, participants will be followed at 6 months of follow-up to assess the occurrence of cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years old admitted to Cardiac Intensive Care Unit (CCU) for any reason.
* Oral informed consent.

Exclusion Criteria:

* Hospitalization for a planned interventional procedure (percutaneous coronary intervention, coronary artery bypass graft surgery, transcatheter aortic valve implantation…).
* Dementia.
* Hospitalization for more than 24 hours at any hospital facility before admission to the CCU.
* Patient under legal protection without the consent of the legal representative.
* Patient with no social security.
* Declining participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients over 18 years admitted to the CCU. The main exclusion criteria will be hospitalization for a planned interventional procedure, dementia, or hospitalization for more than 24 hours at any hospital facility before admission to the CCU. Informed consent will be obtained from all participants.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-06-06 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of psychoactive drug use assessed by urine drug assay at the time of patient admission. | Day 0
  The following psychoactive drugs will be evaluated for all consecutive patients by urine drug assay (NarcoCheck®, Kappa City Biotech SAS, Montluçon, France) within two hours of admission to the CCU: i) cannabinoids (tetrahydrocannabinol [THC]), including cannabis and hashish; ii) cocaine and metabolites, including cocaine and crack; iii) amphetamines; iv) MDMA; and v) heroin and other opioids.
  In addition to the analysis of psychoactive drug use, the investigators will also use the NarcoCheck® urine drug assay to evaluate the associated use of the following psychostimulant drugs: barbiturates, benzodiazepines, tricyclic antidepressant drugs, methadone and buprenorphine.

SECONDARY OUTCOMES:
In-hospital major adverse events (MAE) | Up to 3 months
  In-hospital major adverse events (MAE) will be a combined outcome including:
  * all-cause mortality,
  * cardiogenic shock according to the European Society of Cardiology (ESC) guidelines, and requiring medical (catecholamines or inotropic agents) or mechanical haemodynamic support
  * cardiac arrest: severe ventricular arrhytmia requiring defibrillation or anti-arrhytmic agents
  This outcome will be assessed by the clinical team in charge of the CCU during the hospitalization.
Duration of the hospitalization | Up to 3 months
  The duration of the hospitalization of each patient in CCU and in the hospital.
Combined major adverse clinical events (MACE). | 12 months of follow-up
  MACE will be defined as all-cause death or unplanned hospitalization for acute cardiovascular reasons, confirmed by independent adjudication experts who will review medical documents according to the standardized definitions.
All cause mortality | 12 months of follow-up
  The adjudication of all-cause death was performed using the electronic French National Registry of Death (Institut National de la Statistique et des Etudes Economiques, INSEE registry).
The occurrence of cardiovascular events | 12 months of follow-up
  Other secondary outcomes will be assessed by independent adjudication experts will be as follows: all-cause death, cardiovascular mortality, nonfatal myocardial infarction, unstable angina, resuscitated cardiac arrest, hospitalizations for heart failure, heart transplantation or implantation of a mechanical circulatory support device, sustained ventricular arrhythmias, coronary revascularization, stroke, venous thromboembolic events, endocarditis and the implantation of a pacemaker or implantable cardioverter-defibrillator.
Combined major adverse clinical events (MACE). | 24 months of follow-up
  MACE will be defined as all-cause death or unplanned hospitalization for acute
All cause mortality | 24 months of follow-up
  The adjudication of all-cause death was performed using the electronic French National Registry of Death (Institut National de la Statistique et des Etudes Economiques, INSEE registry).
The occurrence of cardiovascular events | 24 months of follow-up
  Other secondary outcomes will be assessed by independent adjudication experts will be as follows: all-cause death, cardiovascular mortality, nonfatal myocardial infarction, unstable angina, resuscitated cardiac arrest, hospitalizations for heart failure, heart transplantation or implantation of a mechanical circulatory support device, sustained ventricular arrhythmias, coronary revascularization, stroke, venous thromboembolic events, endocarditis and the implantation of a pacemaker or implantable cardioverter-defibrillator.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Guillaume DILLINGER, MD,PhD, Study Director — Lariboisière Hospital, APHP, Paris
Locations (1):
- CHU Lariboisière, APHP, Cardiology, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fauvel C, Dillinger JG, Bochaton T, Levasseur T, El Ouahidi A, Zakine C, El Hadad A, Mansencal N, Noirclerc N, Goralski M, Thuaire C, Mewton N, Schurtz G, Lim P, Pommier T, Lemarchand L, Laissac Q, Lamblin N, Boukertouta T, Logeart D, Cohen-Solal A, Henry P, Pezel T; ADDICT-ICCU Investigators. In-hospital and 1 year incremental prognostic value of drug abuse detection in acute heart failure. ESC Heart Fail. 2025 Aug;12(4):2736-2748. doi: 10.1002/ehf2.15118. Epub 2025 May 21. PMID 40396434
- [Derived] Weizman O, Hamzi K, Henry P, Schurtz G, Hauguel-Moreau M, Trimaille A, Bedossa M, Dib JC, Attou S, Boukertouta T, Boccara F, Pommier T, Lim P, Bochaton T, Millischer D, Merat B, Picard F, Grinberg N, Sulman D, Pasdeloup B, El Ouahidi Y, Goncalves T, Vicaut E, Dillinger JG, Toupin S, Pezel T; ADDICT-ICCU Investigators. Machine learning score to predict in-hospital outcomes in patients hospitalized in cardiac intensive care unit. Eur Heart J Digit Health. 2024 Dec 20;6(2):218-227. doi: 10.1093/ehjdh/ztae098. eCollection 2025 Mar. PMID 40110223
- [Derived] Sibilia B, Toupin S, Bouali N, Brette JB, Ramonatxo A, Schurtz G, Hamzi K, Trimaille A, Gall E, Piliero N, Unger A, Andrieu S, Goncalves T, Picard F, Roule V, Roubille F, Houssany-Pissot S, Bouchot O, Aboyans V, Vasram RR, Bochaton T, Logeart D, Solal AC, Cartailler J, Mebazaa A, Dillinger JG, Henry P, Pezel T. Supervised machine learning including environmental factors to predict in-hospital outcomes in acute heart failure patients. Eur Heart J Digit Health. 2024 Dec 16;6(2):190-199. doi: 10.1093/ehjdh/ztae094. eCollection 2025 Mar. PMID 40110211
- [Derived] Hamzi K, Gall E, Roubille F, Trimaille A, Elbaz M, El Ouahidi A, Noirclerc N, Fard D, Lattuca B, Fauvel C, Goralski M, Alvain S, Chaib A, Piliero N, Schurtz G, Pommier T, Bouleti C, Tron C, Bonnet G, Nhan P, Auvray S, Lequipar A, Dillinger JG, Vicaut E, Henry P, Toupin S, Pezel T; ADDICT-ICCU Investigators. Phenotypic clustering of patients hospitalized in intensive cardiac care units: Insights from the ADDICT-ICCU study. Arch Cardiovasc Dis. 2024 Jun-Jul;117(6-7):392-401. doi: 10.1016/j.acvd.2024.03.004. Epub 2024 May 23. PMID 38834393
- [Derived] Fauvel C, Dillinger JG, Bouleti C, Trimaille A, Tron C, Chaussade AS, Thuaire C, Delmas C, Boccara A, Roule V, Millischer D, Thevenet E, Meune C, Stevenard M, Charbonnel C, Maitre Ballesteros L, Pommier T, El Ouahidi A, Swedsky F, Martinez D, Hauguel-Moreau M, Schurtz G, Coisne A, Dupasquier V, Bochaton T, Gerbaud E, Puymirat E, Henry P, Pezel T; ADDICT-ICCU Investigators. Tricuspid annular plane systolic excursion over systolic pulmonary artery pressure prognostic value for in-hospital adverse events in patients hospitalized for acute coronary syndrome. Eur Heart J Cardiovasc Imaging. 2024 Aug 26;25(9):1244-1254. doi: 10.1093/ehjci/jeae110. PMID 38650518
- [Derived] Fauvel C, Dillinger JG, Rossanaly Vasram R, Bouleti C, Logeart D, Roubille F, Meune C, Ohlmann P, Bonnefoy-Coudraz E, Albert F, Attou S, Boukhris M, Pommier T, Merat B, Noirclerc N, Bouali N, Aghezzaf S, Schurtz G, Mansencal N, Andrieu S, Henry P, Pezel T; ADDICT-ICCU Investigators. In-hospital prognostic value of TAPSE/sPAP in patients hospitalized for acute heart failure. Eur Heart J Cardiovasc Imaging. 2024 Jul 31;25(8):1099-1108. doi: 10.1093/ehjci/jeae059. PMID 38428980
- [Derived] Clement A, Dillinger JG, Ramonatxo A, Roule V, Picard F, Thevenet E, Swedzky F, Hauguel-Moreau M, Sulman D, Stevenard M, Amri N, Martinez D, Maitre-Ballesteros L, Landemaine T, Coppens A, Bouali N, Guiraud-Chaumeil P, Gall E, Lequipar A, Henry P, Pezel T. In-hospital prognosis of acute ST-elevation myocardial infarction in patients with recent recreational drug use. Eur Heart J Acute Cardiovasc Care. 2024 May 7;13(4):324-332. doi: 10.1093/ehjacc/zuae024. PMID 38381068
- [Derived] Dillinger JG, Pezel T, Delmas C, Schurtz G, Trimaille A, Piliero N, Bouleti C, Lattuca B, Andrieu S, Fabre J, Rossanaly Vasram R, Dib JC, Aboyans V, Fauvel C, Roubille F, Gerbaud E, Boccara A, Puymirat E, Toupin S, Vicaut E, Henry P; ADDICT-ICCU trial. Carbon monoxide and prognosis in smokers hospitalised with acute cardiac events: a multicentre, prospective cohort study. EClinicalMedicine. 2024 Jan 3;67:102401. doi: 10.1016/j.eclinm.2023.102401. eCollection 2024 Jan. PMID 38261914
- [Derived] Pezel T, Dillinger JG, Trimaille A, Delmas C, Piliero N, Bouleti C, Pommier T, El Ouahidi A, Andrieu S, Lattuca B, Rossanaly Vasram R, Fard D, Noirclerc N, Bonnet G, Goralski M, Elbaz M, Deney A, Schurtz G, Docq C, Roubille F, Fauvel C, Bochaton T, Aboyans V, Boccara F, Puymirat E, Batisse A, Steg G, Vicaut E, Henry P; ADDICT-ICCU Investigators. Prevalence and impact of recreational drug use in patients with acute cardiovascular events. Heart. 2023 Oct 12;109(21):1608-1616. doi: 10.1136/heartjnl-2023-322520. PMID 37582633